CLINICAL TRIAL: NCT05093998
Title: Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of AV5080 in Patients With Uncomplicated Influenza
Brief Title: Study Evaluating the Efficacy and Safety of AV5080 in Patients With Uncomplicated Influenza
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Viriom (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FLU-AV5080-03
Record Dates: First submitted 2021-10-22; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Influenza
Keywords: Treatment for influenza in adults
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This study is double-blind. Clinical center staff and patients will not know what therapy and in what doses are prescribed for each individual patient. Blinding will be achieved by masking the AV5080/placebo drug (each patient will take a pill corresponding to 80 mg or placebo) and dispensing the drug using IWRS. Each patient will be given the study drug in banks. Banks will have a unique identification number, otherwise they will be identical in marking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1. (Experimental): AV5080 at a daily dose of 160 mg
  Interventions: Drug: AV5080
- Group 2. (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AV5080 — oral hard gelatin capsules
  Other Names: AV5080 at a daily dose of 160 mg
  Arms: Group 1.
Other: Placebo — Hard gelatin capsules with a white body
  Arms: Group 2.

SUMMARY:
To evaluate the efficacy of AV5080 versus Placebo based on time to symptom resolution in patients with uncomplicated influenza.

DETAILED DESCRIPTION:
This study is an international, multicenter, double-blind, randomized, placebo-controlled, phase III clinical trial in parallel groups evaluating the efficacy and safety of AV5080 in patients with uncomplicated influenza.

Only patients with mild to moderate influenza, without complications, will be included in the study. Taking into account the seasonality of the pathology and the low percentage of influenza in the general structure of ARVI incidence, for the successful inclusion of all patients in the study during two epidemiological seasons. The study will enroll 700 patients aged 18 to 65 years with a confirmed clinical diagnosis of influenza to treatment (AV5080) and placebo cohorts (1:1).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Men and women between the ages of 18 and 65 (inclusive).
3. Outpatients (including those admitted at home) and inpatients hospitalized for epidemiological reasons, diagnosed with influenza (ICD 10: J10 Influenza caused by an identified influenza virus) of mild to moderate severity.
4. Positive result of the rapid enzyme immunoassay test for influenza virus at screening.
5. Increase in body temperature in the armpit up to ≥ 38.0 оС at screening (or within 24 hours before screening according to the patient's words).
6. Presence of at least one of the following symptoms of moderate severity on screening:

   headache, weakness/malaise, muscle pain/aches, fever/chills.
7. The duration of the disease is no more than 48 hours at the time of screening according to the patient.
8. Consent of patients to use adequate methods of contraception throughout the study.

Adequate methods of contraception include the use of:

* oral or transdermal contraceptives;
* a condom or diaphragm (barrier method) with spermicide or
* an intrauterine device.

Exclusion Criteria:

1. Pregnant or lactating women or women planning pregnancy during a clinical study; women capable of childbearing (including menopausal women less than 2 years old) who do not use adequate methods of contraception.
2. Individual intolerance to the drug AV5080 or its components. Lactase deficiency, lactose intolerance, glucose-galactose malabsorption.
3. Presence of complications of influenza, signs of bacterial infection or severe flu at the time of screening.
4. Infectious diseases transferred during the last week before screening
5. The need for hospital treatment for influenza, with the exception of hospitalization for epidemiological indications.
6. Reception of neuraminidase inhibitors (zanamivir and oseltamivir), immunotropic drugs, systemic glucocorticosteroids, antibacterial drugs of systemic action within 1 month before screening. Taking drugs that prolong the QT interval on an ECG (quinidine, amiodarone, procainamide, phenothiazine derivatives) for 5 half-lives or less before screening.
7. A history of influenza vaccination within 3 months prior to screening.
8. Chronic diseases of the respiratory system (bronchial asthma, COPD,) in history.
9. Persons with metabolic disorders (diabetes mellitus, obesity of 2-3 degrees).
10. Hypokalemia at screening (potassium level less than 3.5 mmol/L)
11. Persons with chronic kidney disease, chronic liver disease, with certain neurological conditions (including neuromuscular, neurocognitive disorders, epilepsy), hemoglobinopathies or suppressed immune conditions, or due to primary immunosuppressive conditions such as HIV infection, or in connection with secondary immunodeficiency states due to the intake of immunosuppressive medications or malignant neoplasms.
12. Significant cardiovascular diseases at present or during 12 months before screening, including: prolongation of the QT interval on ECG more than 450 ms, atrioventricular block, sinus bradycardia, chronic cerebrovascular insufficiency, chronic heart failure class III or IV (according to the classification of the New York Heart Association), severe arrhythmia, requiring treatment with class Ia, Ib, Ic, or III antiarrhythmic drugs, unstable angina pectoris, myocardial infarction, heart and coronary artery surgery, significant heart valve disease, transient ischemic attack or stroke, uncontrolled hypertension with systolic blood pressure> 180 mm Hg ... and diastolic blood pressure> 110 mm Hg, pulmonary embolism or deep vein thrombosis.
13. A history of chronic alcoholism, drug addiction or dependence on other chemical compounds.
14. Participation in other clinical trials within 3 months prior to screening.
15. Inability to read or write; unwillingness to understand and follow research protocol procedures; non-compliance with the regimen of taking medications or performing procedures that, in the opinion of the Investigator, may affect the results of the study or the safety of the patient and prevent the patient from further participation in the study any other comorbid medical or serious mental condition that renders a patient ineligible for participation in a clinical research study, limits the ability to obtain informed consent, or may affect a patient's ability to participate in a study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2022-01-15 (Estimated); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Time to symptom resolution | 30 days
  The resolution of influenza symptoms is confirmed by the absence of symptoms or their reduction to mild severity (0-1 points) and a decrease in body temperature in the armpit to ≤ 37.2 °C for at least 24 hours. The time to resolve the flu symptoms is the start time of the 24-hour (or longer) interval.

SECONDARY OUTCOMES:
Profile of changes in influenza virus titer versus time (AUC) for 192 hours (in inpatients) | 192 hours
Frequency of symptom resolution within 96 hours of initiation of study therapy | 96 hours
Frequency of elimination of influenza virus before Day 6 | 6 Days
The incidence of complications from influenza | 30 days

CONTACTS AND LOCATIONS:
Locations (6):
- Russia (6):
  - Specialized Clinical Infectious Diseases Hospital, Krasnodar
  - Murmansk Regional Clinic named after P.A. Bayandin, Murmansk
  - Federal Research Center Institute of Cytology and Genetics, Siberian Branch of the Russian Academy of Sciences, Novosibirsk
  - Center for the Prevention and Control of AIDS and Infectious Diseases, Saint Petersburg
  - First Saint Petersburg State Medical University named after I.I. Academician Pavlov, Saint Petersburg
  - Research Center Eco-safety, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No